CLINICAL TRIAL: NCT02319252
Title: Gastric- Versus Jejunal Feeding Tubes in Alcoholic Liver Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tubes in liver diseases
Record Dates: First submitted 2014-12-02; First posted 2014-12-18 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2016-05

CONDITIONS: Malnutrition; Liver Diseases, Alcoholic
MeSH Terms: conditions — Malnutrition; Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastric tube (Active Comparator): A gastric tube is used
  Interventions: Device: Gastric tube (Nutricia Flocare® Pur Tube Enlock)
- Jejunal tube (Active Comparator): A jejunal tube is used
  Interventions: Device: Jejunal tube (Nutricia Flocare® Bengmark®)

INTERVENTIONS:
Device: Gastric tube (Nutricia Flocare® Pur Tube Enlock) — Nutricia Flocare® Pur Tube Enlock, Ch. 12
  Arms: Gastric tube
Device: Jejunal tube (Nutricia Flocare® Bengmark®) — Nutricia Flocare® Bengmark®, Ch. 10
  Arms: Jejunal tube

SUMMARY:
The study is an unblinded randomized trial, designed to examine whether gastric- or jejunal feeding tubes are the most effect full to feed patients with alcoholic liver diseases and non-sufficient oral intake.

The primary outcome will be differences in nutrition intake between the groups. Secondary outcomes will be: the amount of unplanned tube discontinuations; handgrip and patients' quality of life, nausea & vomiting.

The study will include 40 patients at Aarhus University Hospital, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic liver disease
* nutrition intake less than 75% of needed intake
* Signed informed consent form

Exclusion Criteria:

* Hepatic encephalopathy, grade 3 - 4
* Anatomic barriers to have a tube placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Differences in nutrition intake | Day 3 & 7 and every 7th. day until discharge from the hospital, up to 3 months
  Nutrition intake, protein intake, oral intake versus tube intake

SECONDARY OUTCOMES:
Differences in patients reported outcomes | Day 3 & 7 and every 7th. day until discharge from the hospital, up to 3 months
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Palle Bager, PhD, Principal Investigator — Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Central Region, Denmark